CLINICAL TRIAL: NCT05838729
Title: Phase 1b/2a Study of RiMO-301 and Hypofractionated Radiotherapy With A PD-1 Inhibitor for the Treatment of Unresectable, Recurrent or Metastatic Head-Neck Cancer
Brief Title: Study of RiMO-301 and Radiotherapy With PD-1 Inhibitor for the Treatment of Head-Neck Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Coordination Pharmaceuticals, Inc. (Industry)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RiMO-HNC-IO1
Record Dates: First submitted 2023-04-13; First posted 2023-05-01 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Head Neck Cancer; Intratumoral Injection
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RiMO-301 (Experimental): Intratumoral injection of RiMO-301 followed by pembrolizumab or nivolumab followed by hypofractionated radiation
  Interventions: Drug: RiMO-301

INTERVENTIONS:
Drug: RiMO-301 — A single dose of RiMO-301 will be administered via an intratumoral injection.
  PD-1 inhibitor (pembrolizumab or nivolumab) will be administered via a 30-minute intravenous infusion until disease progression or unacceptable toxicity.
  Patients will receive hypofractionated radiation in 5 fractions.

SUMMARY:
This is a prospective, open-label, single arm, non-randomized study of RiMO-301 with hypofractionated radiation and a PD-1 Inhibitor in patients with unresectable, recurrent or metastatic head-neck cancer.

DETAILED DESCRIPTION:
Primary Objectives:

* To determine the tolerability of RiMO-301 with hypofractionated X-ray radiotherapy and a PD-1 inhibitor (pembrolizumab or nivolumab) in patients with unresectable, recurrent or metastatic head-neck cancer
* To determine the efficacy of RiMO-301 with hypofractionated X-ray radiotherapy and a PD-1 inhibitor (pembrolizumab or nivolumab)

Secondary Objectives:

* To evaluate progression-free survival for up to 12 months
* To determine overall survival for up to 24 months
* To assess patient quality of life

The target population is patients with unresectable, recurrent or metastatic head-neck cancer which is clinically accessible to intratumoral injection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of head-neck cancer that requires palliative radiotherapy
* Patients with unresectable, recurrent or metastatic HNSCC, regardless if the patients have progressed on or are intolerant to platinum-based chemotherapy prior to study enrollment or if the patients are receiving pembrolizumab in the first line:

  * receiving a PD-1 inhibitor (pembrolizumab or nivolumab) as a standard of care, or
  * suitable to receive a PD-1 inhibitor (pembrolizumab or nivolumab) as a standard of care in the discretion of the treating physician or Principal Investigator
* Must have at least 1 target lesion that is clinically accessible to RiMO-301 injection and amenable to receive RT regimens specified in this protocol
* The selected target lesions must be measurable on cross-sectional imaging and repeated measurements at the same location should be achievable
* Target tumor not in the previously irradiated field or in the field irradiated at least six months prior to RiMO-301 injection and with no complications from the prior radiation course
* RiMO-301 injection to multiple lesions (≤ 5 in total) in a single patient is allowed as long as the total tumor volume does not exceed 250 cm3
* Patient must have recovered from acute toxic effects (≤ grade 1 CTCAEv5) of previous cancer treatments prior to enrollment
* Have adequate bone marrow reserve and adequate liver function
* Have a life expectancy of at least 12 weeks
* ECOG score of 0-2
* Age 18 years or older

Exclusion Criteria:

* Have signs or symptoms of end organ failure, major chronic illnesses other than cancer, or any severe concomitant conditions
* Symptomatic central nervous system metastases and/or carcinomatous meningitis
* Active autoimmune disease that has required systemic treatment in the past 2 years
* Ongoing clinically significant infection at or near the incident lesion
* Major surgery over the target area (excluding placement of vascular access) ≤21 days from beginning of the study drug or minor surgical procedures ≤7 days. No waiting is required following implantable port, enteral feeding tube and catheter placement
* Has received any approved or investigational anti-neoplastic agent or immunotherapy other than PD-1 inhibitors (pembrolizumab or nivolumab) within 4 weeks prior to RiMO-301 injection
* Patients with lesions which have significant blood vessel involvement (such as carotid artery encasement) or other major structures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Determination of Recommended Dose | 6 weeks
  • The dose limiting toxicities of RiMO-301 with hypofractionated X-ray radiotherapy and a PD-1 inhibitor, as assessed by CTCAEv5, will not be observed in 33% or more patients
Evaluation of Anti-Tumor Response | 12 months
  • To determine the objective response rate: complete or partial response, as defined by RECIST and itRECIST

SECONDARY OUTCOMES:
Evaluation of Progression-Free Survival | 12 months
  Time from enrollment to local-regional recurrence, local-regional progression, distant progression or death from any cause, whichever occurs first
Evaluation of Overall Survival | 24 months
  Time from enrollment to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Feldman, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No